CLINICAL TRIAL: NCT01075750
Title: Perioperative Fluid Management in Patients Receiving Cadaveric Renal Transplants - Effects of Normal Saline Versus Balanced Infusates on the Incidence of Electrolyte and Acid-base Disturbances
Brief Title: Perioperative Fluid Management in Patients Receiving Cadaveric Renal Transplants
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Eva Meitner, M.D., Medical University of Vienna
Other Study IDs: MUViennaAnemev
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Hyperkalaemia Requiring Postoperative Dialysis; Metabolic Acidosis
Keywords: hyperkalaemia; metabolic acidosis; renal transplantation; normal saline; elomel isoton; fluid management in renal transplantation
MeSH Terms: conditions — Acidosis; Hyperkalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal Saline: Patients receiving Normal Saline during and after the renal transplantation.
- Elomel Isoton: Patients receiving Elomel Isoton during and after renal transplantation

SUMMARY:
In this study we want to show that the choice of a balanced type fluid solution for the perioperative fluid management of patients receiving cadaveric renal transplantation results in less occurrence of intra- and postoperative hyperkalemia, and thus the need for postoperative dialysis. Additionally, we aim to determine whether the use of a balanced infusion solution leads to less occurrence of metabolic acidosis and electrolyte disorders than the use of isotonic saline.

Furthermore we want to evaluate whether perioperative fluid management with balanced infusion solutions results in a higher frequency of primary graft function than with administration of isotonic saline.

We will test the hypothesis that the use of "Elomel isoton"(Fresenius Kabi Austria GmbH) a balanced infusion solution will result in less occurrence of hyperkalemia and consequent post-transplant dialysis, less occurrence of metabolic acidosis, decreased incidence of electrolyte disorders and higher incidence of primary graft function when compared to isotonic saline for perioperative fluid management in patients receiving cadaveric renal transplantation.

DETAILED DESCRIPTION:
Background

Kidney transplantation is the treatment of choice for patients with end-stage-renal-disease (ESRD). Successful renal transplantation improves quality of life and reduces mortality in eligible patients when compared to hemodialysis. In 2007, 44 kidney transplantations per million residents were performed in Austria. The number of patients with a renal transplant has continuously risen in the last ten years. 398 kidney transplantations were performed in Austria in 2007, of which only 61 were of living donors. This underlines the special role of cadaveric kidney transplantation in Austria.

Several studies have demonstrated that adequate intraoperative fluid administration is associated with earlier onset of graft function and improved graft survival in renal transplant recipients. However, which kind of solution should be chosen for the perioperative fluid management of renal transplant recipients remains to be clarified. A non-governmental US survey has shown that normal saline is the most commonly used fluid for renal transplantation. The most common cited reason for the administration of normal saline was the lack of potassium in the solution. Balanced salt type fluids were used in only less than 10% of kidney transplantations.

To our knowledge only three studies compared the effects of lactated ringer's solution versus normal saline in kidney transplantation. Taken together, the application of lactated ringer's solution led to less occurrence of metabolic acidosis, electrolyte derangements and in one study, the appearance of hyperkalemia was eliminated by the use of lactated ringer's instead of normal saline. However, it was also shown that the administration of lactated ringer's during kidney transplantation led to a significant rise in lactate levels compared to those treated with normal salin. Despite the knowledge that lactated ringer's can at least potentially lead to a rise in lactate levels, no studies using acetate based balanced salt type fluids have been performed so far in cadaveric renal transplantation. We therefore propose a prospective study in which patients undergoing cadaveric kidney transplantation will be randomized to receive either a solely acetate buffered balanced salt type fluid or a normal saline for infusion therapy.

Clinical considerations

Postoperative hyperkalemia is a common problem in patients receiving cadaveric renal transplantation, especially when primary graft function does not occur. Due to the acidifying effect of isotonic saline infusion via the generation of hyperchloremic acidosis and/or dilutional acidosis, a rise in serum potassium is only boosted. However, today isotonic saline is the most commonly used infusion solution for the perioperative period in renal transplantation.

The use of a balanced infusion solution, containing a metabolizable anion, such as acetate, could result in less metabolic acidosis and therefore a decreased need for post-transplant dialysis. Moreover, since balanced infusion solutions have a by far lower chloride content than isotonic saline, the adverse effects of a rise in serum chloride on renal perfusion could be avoided. This could ultimately result in improved graft function.

Preliminary studies

O'Malley et al. compared the effects of lactated Ringer's to isotonic saline in 51 renal transplant patients. 48 patients received living donor transplantation and 3 received cadaveric renal transplantation. 26 patients received isotonic saline and 25 lactated Ringer's. 19% of patients receiving isotonic saline reached postassium concentrations > 6mmol/L and required treatment versus 0% in the lactated Ringer's group. 31% of patients in the isotonic saline group versus 0% in the lactated Ringer's group required treatment for metabolic acidosis. No effect on primary graft function could be shown.

Hadimioglu et al. randomized patients undergoing living-related kidney transplantation to three groups receiving either isotonic saline, lactated Ringer's or Plasmalyte (a balanced infusion solution using acetate and gluconate). No effects on potassium levels could be shown in this study. Patients receiving isotonic saline showed significant decreases in pH, base excess and a significant rises in serum chloride. In the lactated Ringer's group lactate levels increased significantly. The study showed no differences in the need for postoperative dialysis.

Khajavi et al. randomized patients undergoing kidney transplantation to either normal saline or lactated Ringer's. The authors noticed a higher incidence of hyperkalemia and acidosis in the isotonic saline group while 2 patients in the lactated Ringer's group lost their kidneys due to vascular graft thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* All patients with end-stage-renal disease admitted for cadaveric renal transplantation will be included in the study

Exclusion Criteria:

* Patients younger than 18 years of age
* Hyperkalemia defined as a serum potassium exceeding 5.5 mmol/L pre-operatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving a cadaveric renal transplant in the General Hospital of Vienna
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
intra or postoperative hyperkalaemia | 7 days

SECONDARY OUTCOMES:
metabolic acidosis | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Edith Fleischmann, Univ.Prof, Study Chair — Medical University of Vienna; Gregor Lindner, MD, Study Director — Inselspital Bern, University of Bern; Eva Meitner, MD, Principal Investigator — Medical University of Vienna; Peter Biesenbach, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna/General Hospital of Vienna, Vienna, Vienna, Austria